CLINICAL TRIAL: NCT03918759
Title: Diagnostic Accuracy of 68Gallium Positron Emission Tomography/ Magnetic Resonance Imaging (68Ga PET/MRI), Endoscopic Ultrasound (EUS) and Computed Tomography in the Assessment of Lymph Node Metastases by Nonfunctioning Pancreatic Neuroendocrine Neoplasms
Brief Title: Diagnostic Accuracy of Preoperative Diagnostic Procedure in the Assessment of Lymph Node Metastases by NF-PanNENs
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Massimo Falconi, Principal Investigator, IRCCS San Raffaele
Other Study IDs: DETECTYON study
Record Dates: First submitted 2018-12-12; First posted 2019-04-18 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Non Functioning Pancreatic Endocrine Tumor
Keywords: Lymph node metastases; Diagnostic accuracy
MeSH Terms: conditions — Non functioning pancreatic endocrine tumor; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pancreatic Neuroendocrine Neoplasms (PanNEN) are a heterogeneous group of neoplasms that arise from the endocrine cells of the pancreatic gland. Non-functioning (NF-PanNEN) represents the most common forms and do not produce syndromes due to hormonal hypersecretion. Several prognostic factors have been demonstrated for NF-PanNEN. The presence of nodal metastasis and lymph node ratio are widely considered predictors of disease-free survival and even the number of positive nodes has been found to be associated with recurrence. In addition to traditional imaging exams, diagnostic work-up should include a Positron Emission Tomography/CT with 68Ga labeled somatostatin analogues, which have shown a high sensitivity and specificity while 18F-FDG PET can be associated for evaluating the possible presence of a high-grade component. Moreover, pancreatic endoscopic ultrasound (EUS) is usually part of the preoperative staging both for imaging details and cytological sampling. Therefore an accurate identification of nodal metastases preoperatively may have important implications for the extent of surgical resection and lymphadenectomy and even for a prognostic outcome.

In this study the investigators will evaluate prospectively the accuracy of these diagnostic exams in detecting the lymph node status. Patients with sporadic NF-PanNEN who are candidates for surgical resection will undergo CE-CT scan, 68Ga DOTATOC (and eventually 18F-FDG) PET/MRI and EUS with FNA/B. Reference standard for defining the presence of nodal metastases is represented by pathological examination on the specimen.

DETAILED DESCRIPTION:
The study is designed as a prospective monocentric observational cohort study. The primary endpoint of the study is to assess the accuracy of preoperative diagnostic procedures in terms of sensitivity and specificity in detecting nodal metastases in sporadic NF-PanNEN as determined by pathological examination on the specimen.

Patients with a suspect of a sporadic NF-PanNEN will be considered for the study at the time of the first visit. All consecutive patients who will meet inclusion criteria, after informed consent, will be included. The preoperative work-up will be performed in our center. All the examinations required for this study are necessary for the correct preoperative staging, representing the standard diagnostic work-up in patients with PanNEN. Computed tomography (CT) images will be obtained by multiphase technique. Non-enhanced, arterial and portal phase images will be obtained in all the patients. Computed tomography (CT) images will be obtained by multiphase technique. Non-enhanced, late arterial and portal phase images will be obtained in all the patients as well. Every lymph nodal finding with short-axis diameter >1cm or with pathological contrast enhancement will be considered as pathological. Pancreatic endoscopic ultrasound (EUS) is a relatively recent endoscopic technique which combines the high-frequency ultrasound technology with the direct endoscopic vision, permitting a sensitive evaluation of pancreatic lesions (from the stomach or the duodenum), an accurate vascular staging and the assessment of pathologic lymph nodes related to the tumor. Nodes larger than 1 cm, with well demarked and/or rounded margins and with typical echoic/elastographic features will be reported as metastatic. Moreover, the additive value of EUS is the possibility to sample pancreatic masses and lymph nodes with a fine needle aspiration (FNA), to obtain a cytological diagnosis. A PET/MRI with 68Ga-DOTATOC is also necessary for the staging of the disease. A 18F-FDG PET will be performed according to the clinician's discretion, especially in the presence of large lesions and/or liver metastases.

As soon as the preoperative assessment will be completed, a surgical resection will be proposed to the patient according to the international guidelines on the management of NF-PanNEN. A standard pancreatic resection will be performed according to the site and the extension of the lesion. Nodes will be classified according to the Japanese classification of the biliary tract cancers. The extension of lymphadenectomy will be related to the type of pancreatic resection.

LN that will be resected apart from the pancreatic specimen, will be sent for pathological examination in a separated cup labelled by the surgeon. In case of preoperative detection of nodal involvement in a station not included in the standard lymphadenectomy, the nodes in this station will be resected to confirm or not the radiological finding. Reference standard for defining the presence of nodal metastases will be represented by the pathological examination.

All data regarding the clinical aspect, the radiological reports and the pathological exam will be fully available only to the surgeon. Radiologist, nuclear medicine physician, and pathologist will be blinded to the radiological findings.

Several retrospective studies 11-12 reported a prevalence of nodal metastases in PanNEN of about 40%, in case of tumors > 2 cm. No data have been found on the sensitivity and specificity of the various examinations in detecting nodal involvement. Given this prevalence and assuming a good accuracy based on this institute experience, the simple size required to assess the sensitivity and specificity of the methods was found to be of 150 patients, considering a 95% confidence interval with a margin of error of 10%.

A descriptive analysis will be performed of the data obtained. The aim will be to evaluate the sensitivity, the specificity and the positive and negative predictive values of the preoperative staging (CE-CT scan, EUS, 68Ga DOTATOC/18F-FDG PET/MRI). The comparison between the exams in terms of prediction of the nodal status will be calculated with the McNemar test. A logistic regression model will be used to assess the risk of nodal positivity at the pathological report when the preoperative imaging demonstrates the features of nodal metastases. OR and 95% confidence interval will be calculated. The statistical correlation between the risk of nodal positivity at the pathological report and some preoperative variables will be evaluated with the chi-square test and ROC curves analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Individuals with a diagnosis of NF-PanNEN undergoing standard pancreatic resection (pancreatoduodenectomy, left pancreatectomy, total pancreatectomy)
* Cytologically/histologically proven diagnosis of NF-PanNEN.
* Informed consent

Exclusion Criteria:

* Age < 18 years
* Absence of cytological/histological confirmation
* Presence of functioning PanNEN
* Presence of genetic syndrome (MEN1, VHL, NF)
* Patients undergone previously to an EUS in another institution with a FNA/B positive for NET

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients with a suspect of a sporadic NF-PanNEN will be considered for the study at the time of the first visit. All consecutive patients who will meet inclusion criteria, after informed consent, will be included. The enrollment will be completed only after the cytological/histological confirmation NF-PanNEN.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of preoperative staging in detecting nodal metastases by evaluating and comparing sensitivity and specificity of the diagnostic techniques | 2 years
  The primary endpoint of the study is to assess the accuracy of preoperative diagnostic procedures in terms of sensitivity and specificity in detecting nodal metastases in sporadic NF-PanNEN

SECONDARY OUTCOMES:
Evaluate the prognostic role of the nodal involvement | 5 years
  The secondary outcomes include the assessment of the prognostic role of nodal involvement on disease/progression free survival in patients who undergo a pancreatic resection for a Non-functioning Pancreatic Neoplasms.
Evaluate the correlation between preoperative radiological and/or clinical data and nodal involvement | 5 years
  This secondary outcome include the evaluation of other possible variables that can be associated with the risk of nodal metastases such as preoperative dimension in mm of the PanNEN, location, features at the imaging, standard uptake value (SUV).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Partelli, MD, PhD, Study Director — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boninsegna L, Panzuto F, Partelli S, Capelli P, Delle Fave G, Bettini R, Pederzoli P, Scarpa A, Falconi M. Malignant pancreatic neuroendocrine tumour: lymph node ratio and Ki67 are predictors of recurrence after curative resections. Eur J Cancer. 2012 Jul;48(11):1608-15. doi: 10.1016/j.ejca.2011.10.030. Epub 2011 Nov 28. PMID 22129889
- [Background] Hashim YM, Trinkaus KM, Linehan DC, Strasberg SS, Fields RC, Cao D, Hawkins WG. Regional lymphadenectomy is indicated in the surgical treatment of pancreatic neuroendocrine tumors (PNETs). Ann Surg. 2014 Feb;259(2):197-203. doi: 10.1097/SLA.0000000000000348. PMID 24253141
- [Background] Partelli S, Javed AA, Andreasi V, He J, Muffatti F, Weiss MJ, Sessa F, La Rosa S, Doglioni C, Zamboni G, Wolfgang CL, Falconi M. The number of positive nodes accurately predicts recurrence after pancreaticoduodenectomy for nonfunctioning neuroendocrine neoplasms. Eur J Surg Oncol. 2018 Jun;44(6):778-783. doi: 10.1016/j.ejso.2018.03.005. Epub 2018 Mar 17. PMID 29610023
- [Background] Deppen SA, Blume J, Bobbey AJ, Shah C, Graham MM, Lee P, Delbeke D, Walker RC. 68Ga-DOTATATE Compared with 111In-DTPA-Octreotide and Conventional Imaging for Pulmonary and Gastroenteropancreatic Neuroendocrine Tumors: A Systematic Review and Meta-Analysis. J Nucl Med. 2016 Jun;57(6):872-8. doi: 10.2967/jnumed.115.165803. Epub 2016 Jan 14. PMID 26769864
- [Background] Miyazaki M, Ohtsuka M, Miyakawa S, Nagino M, Yamamoto M, Kokudo N, Sano K, Endo I, Unno M, Chijiiwa K, Horiguchi A, Kinoshita H, Oka M, Kubota K, Sugiyama M, Uemoto S, Shimada M, Suzuki Y, Inui K, Tazuma S, Furuse J, Yanagisawa A, Nakanuma Y, Kijima H, Takada T. Classification of biliary tract cancers established by the Japanese Society of Hepato-Biliary-Pancreatic Surgery: 3(rd) English edition. J Hepatobiliary Pancreat Sci. 2015 Mar;22(3):181-96. doi: 10.1002/jhbp.211. Epub 2015 Feb 17. PMID 25691463
- [Background] Toste PA, Kadera BE, Tatishchev SF, Dawson DW, Clerkin BM, Muthusamy R, Watson R, Tomlinson JS, Hines OJ, Reber HA, Donahue TR. Nonfunctional pancreatic neuroendocrine tumors <2 cm on preoperative imaging are associated with a low incidence of nodal metastasis and an excellent overall survival. J Gastrointest Surg. 2013 Dec;17(12):2105-13. doi: 10.1007/s11605-013-2360-9. Epub 2013 Oct 8. PMID 24101447
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Result] Dasari A, Shen C, Halperin D, Zhao B, Zhou S, Xu Y, Shih T, Yao JC. Trends in the Incidence, Prevalence, and Survival Outcomes in Patients With Neuroendocrine Tumors in the United States. JAMA Oncol. 2017 Oct 1;3(10):1335-1342. doi: 10.1001/jamaoncol.2017.0589. PMID 28448665
- [Result] Gao Y, Gao H, Wang G, Yin L, Xu W, Peng Y, Wu J, Jiang K, Miao Y. A meta-analysis of Prognostic factor of Pancreatic neuroendocrine neoplasms. Sci Rep. 2018 May 8;8(1):7271. doi: 10.1038/s41598-018-24072-0. PMID 29739948
- [Derived] Partelli S, Muffatti F, Andreasi V, Giannone F, Rossi G, Palumbo D, Mapelli P, Schiavo Lena M, Arcidiacono PG, De Cobelli F, Picchio M, Doglioni C, Falconi M. A Single-center Prospective Observational Study Investigating the Accuracy of Preoperative Diagnostic Procedures in the Assessment of Lymph Node Metastases in Nonfunctioning Pancreatic Neuroendocrine Tumors. Ann Surg. 2022 Nov 1;276(5):921-928. doi: 10.1097/SLA.0000000000005615. Epub 2022 Aug 5. PMID 35930017